CLINICAL TRIAL: NCT00473876
Title: Metformin in Insulin Resistant LV Dysfunction, a Double-blind, Placebo-controlled Trial (TAYSIDE Trial)
Brief Title: Metformin in Insulin Resistant Left Ventricular (LV) Dysfunction (TAYSIDE Trial)
Acronym: TAYSIDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Aaron K Wong, Doctor, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WON001
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Results first posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-05

CONDITIONS: Congestive Heart Failure; Insulin Resistance
Keywords: Chronic Heart Failure; Insulin Resistance; Metformin; Peak VO2
MeSH Terms: conditions — Heart Failure; Insulin Resistance | interventions — Metformin; Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Receiving Metformin for 4 months
  Interventions: Drug: Metformin
- 2 (Placebo Comparator): Matched Placebo for 4 months
  Interventions: Drug: Matched Placebo (Capsules)

INTERVENTIONS:
Drug: Metformin — Started at 500mg bd for 2 weeks. If well tolerated, increase to 1000mg bd for 14 weeks
  Arms: 1
Drug: Matched Placebo (Capsules) — Similar dosing regime as active comparator
  Arms: 2

SUMMARY:
Will metformin improve exercise capacity in chronic heart failure patients who has insulin resistance (pre-diabetic- means before they become diabetic)?

DETAILED DESCRIPTION:
Exercise incapacity is one of the major debilitating symptoms of heart failure patients. Studies showed that heart failure patients will become insulin resistance (IR) or vice versa, severity of heart failure also correlates with the severity of insulin resistance. A recent study demonstrated that if we correct diabetic patient insulin resistance by giving them a drug to make them more sensitive to the effects of insulin, their exercise capacity improves. Therefore, we think that the same effects might happen in heart failure patients who have been identified to the insulin resistance by blood test. Insulin resistance means that they have not yet become diabetic and it is a stage the diabetic patients go through before they develop diabetes.

Therefore, we plan to use a drug called metformin (a diabetic drug), give it to heart failure patients who also have IR for 4 months and examine the effects before and after 4 months of treatment. It is a double blind control study, therefore, neither the examiner nor the patient know which drug they receive (either active drug- Metformin, or a placebo).

The main objective is to assess their exercise capacity using an exercise test called Innocor System. It is a bicycle based exercise test that involves patient breathing into a mouth piece before and during exercise in order for the machine to work out the maximum oxygen consumption and pumping power of the heart.

The other objectives of the trial are looking at the possible mechanisms of improving exercise capacity. We aim to answer the following questions by doing the following tests:

Does exercise capacity improve because of

1. The effect of metformin on the heart? We will answer this question by doing an ultrasound scan of the heart (Echocardiography)
2. The effects on the blood vessels? We plan to perform a test called flow-mediated dilatation, it is an ultrasound scan of the artery in the arm and also assess the blood flow in the skin using a test called Laser Doppler scan (small amount of medication will be delivered through a small electric current and the blood vessels response will be assessed using the laser doppler scan)
3. The effects on the muscle? We will do a muscle biopsy looking at the enzymes activities in the muscle before and after taking 4 months of medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 25-80 yrs with compensated CHF in NYHA functional I-III with evidence of insulin resistance [fasting insulin resistance index values of > 2.7 are said to have insulin resistance].
* Documented Left ventricular systolic dysfunction or LV ejection fraction < 35%

Exclusion Criteria:

* Elderly patients (aged >80 yrs);
* Patients with decompensated CHF (NYHA functional class IV and /or signs of decompensated CHF);
* Renal dysfunction (serum creatinine > 160 mmol/L);
* Patients who are unable to exercise including patients that will be excluded for reasons of safety or potential effects on exercise performance. Therefore, patients with angina or other cardiac or pulmonary symptoms potentially limiting exercise performance will be excluded.
* Systolic blood pressure >190 mmHg at rest or >250 mmHg with exercise or diastolic blood pressure >95 mmHg at rest or >105 mmHg with exercise will also be a reason for exclusion;
* Patients with underlying disease likely to limit life span and/or increase risk of interventions will be excluded i.e., cancer; cardiovascular disease .i.e., uncontrolled hypertension: SBP>180 mmHg or DBP, recent stroke, any severe chronic disease (including renal and hepatic disease).

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chim Lang, MD, FRCP, Principal Investigator — University of Dundee, Scotland
Locations (1):
- Medicine and Therapeutics, Ninewells Hospital, Dundee, Scotland, United Kingdom

REFERENCES:
- [Derived] Schiavone M, Gasperetti A, Vogler J, Compagnucci P, Laredo M, Breitenstein A, Gulletta S, Martinek M, Kaiser L, Tundo F, Palmisano P, Rovaris G, Curnis A, Kuschyk J, Biffi M, Tilz R, Di Biase L, Tondo C, Forleo GB; i-SUSI investigators. Sex differences among subcutaneous implantable cardioverter-defibrillator recipients: a propensity-matched, multicentre, international analysis from the i-SUSI project. Europace. 2024 May 2;26(5):euae115. doi: 10.1093/europace/euae115. PMID 38696701
- [Derived] Schiavone M, Gasperetti A, Compagnucci P, Vogler J, Laredo M, Montemerlo E, Gulletta S, Breitenstein A, Ziacchi M, Martinek M, Casella M, Palmisano P, Kaiser L, Lavalle C, Calo L, Seidl S, Saguner AM, Rovaris G, Kuschyk J, Biffi M, Di Biase L, Dello Russo A, Tondo C, Della Bella P, Tilz R, Forleo GB; iSUSI investigators. Impact of ventricular tachycardia ablation in subcutaneous implantable cardioverter defibrillator carriers: a multicentre, international analysis from the iSUSI project. Europace. 2024 Mar 30;26(4):euae066. doi: 10.1093/europace/euae066. PMID 38584394
- [Derived] Gasperetti A, Schiavone M, Ziacchi M, Vogler J, Breitenstein A, Laredo M, Palmisano P, Ricciardi D, Mitacchione G, Compagnucci P, Bisignani A, Angeletti A, Casella M, Picarelli F, Fink T, Kaiser L, Hakmi S, Calo L, Pignalberi C, Santini L, Lavalle C, Pisano E, Olivotto I, Tondo C, Curnis A, Dello Russo A, Badenco N, Steffel J, Love CJ, Tilz R, Forleo G, Biffi M. Long-term complications in patients implanted with subcutaneous implantable cardioverter-defibrillators: Real-world data from the extended ELISIR experience. Heart Rhythm. 2021 Dec;18(12):2050-2058. doi: 10.1016/j.hrthm.2021.07.008. Epub 2021 Jul 14. PMID 34271173
- [Derived] Cameron AR, Morrison VL, Levin D, Mohan M, Forteath C, Beall C, McNeilly AD, Balfour DJ, Savinko T, Wong AK, Viollet B, Sakamoto K, Fagerholm SC, Foretz M, Lang CC, Rena G. Anti-Inflammatory Effects of Metformin Irrespective of Diabetes Status. Circ Res. 2016 Aug 19;119(5):652-65. doi: 10.1161/CIRCRESAHA.116.308445. Epub 2016 Jul 14. PMID 27418629
- [Derived] Wong AK, Symon R, AlZadjali MA, Ang DS, Ogston S, Choy A, Petrie JR, Struthers AD, Lang CC. The effect of metformin on insulin resistance and exercise parameters in patients with heart failure. Eur J Heart Fail. 2012 Nov;14(11):1303-10. doi: 10.1093/eurjhf/hfs106. Epub 2012 Jun 27. PMID 22740509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with symptomatic CHF were recruited from out patient cardiology clinics and local echocardiography database. Eligible patients were approached to have a fasting blood test to determine their fasting insulin resistance index (FIRI). CHF patients with a FIRI >2.7 were considered to have IR and invited to participate in the study.
Pre-assignment Details: 127 patients were invited for screening.53 patients were excluded based on exclusion criteria.12 patients decided not to continue with the study after screening.62 patients were randomised using a computer generated sequence.Metformin was started at lower dose of 500mg bd for 2 weeks. Doses were up titrated if well tolerated to the target dose.
Groups:
- Metformin: Receiving Metformin for 4 months with a target dose of 1000mg twice a day
- Placebo: Matched Placebo for 4 months
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 39 | 23
Completed | 36 | 22
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 39 | 23 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 9 | 32
  >=65 years | 16 | 14 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (8) | 68 (7) | 65 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 35 | 22 | 57
Region of Enrollment [Number; unit: participants]
  United Kingdom | 39 | 23 | 62

OUTCOME MEASURES:

1. Primary Outcome: Peak VO2
Description: Peak VO2 after 4 months of intervention with either metformin or placebo. The Mean difference between baseline and after 4 months was analyzed using t-test comparing metformin and placebo.
Time Frame: 4 months
Population: .In the metformin group,3 patients were lost to follow up therefore excluded from analysis.5 patients were discontinued on medications due to side effects, however,were included in our intention to treat analysis.In the placebo group,1 patient was lost to follow up and was excluded from analysis
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- Metformin Arm: Peak VO2 mean difference between baseline and after 4 months of metformin was analysed
- Placebo: Peak VO2 mean difference between baseline and after 4 months of placebo
Arm/Group | Metformin Arm | Placebo
Number analyzed (Participants) | 36 | 22
ml/kg/min | -0.38 (1.4) | 3.6 (3.9)
Statistical Analysis 1: Comparison: Metformin Arm vs Placebo; Null hypothesis: Metformin has no effect on peak VO2. We targetted 66 subjects and power calculation based on our previous observational study of CHF with insulin resistance with mean peak VO2 of 11; Test type: Superiority or Other; p = 0.08, t-test, 1 sided; The differences between baseline and post-intervention (4 months) was analyzed using independent t-test, comparing metformin and placebo; Mean Difference (Net) = -0.38

2. Secondary Outcome: Possible Mechanisms That Can Explain the Improvement of Exercise Capacity
Description: VE/VCO2 Slope, measurement of the abnormal ventilatory response to exercise identified by an increased slope of ventilation (L/min) vs. CO2 production (VE/VCO2) (L/min) to incremental workload
Time Frame: 4 months
Population: 39 patients were randomized with 3 dropped out. Therefore, 36 were included in the analysis. There was 1 patient who dropped out in the placebo arm and hence 22 patients were analysed.
Measure: Mean (Standard Deviation); unit: Unitless
Groups:
- Metformin Arm: Assess impact of metformin on submaximal exercise parameters- VE/VCO2 slope (pre-specified end point). The mean VE/VCO2 difference was compared between baseline and after 4 months of metformin.
- Placebo: Impact of placebo on VE/VCO2 slope.
Arm/Group | Metformin Arm | Placebo
Number analyzed (Participants) | 36 | 22
Unitless | -4.45 (10.72) | -0.23 (3.54)
Statistical Analysis 1: Comparison: Metformin Arm vs Placebo; Null hypothesis: Metformin has no effect on the ratio between VCO2 (production of CO2) and VE (ventilation), it is also called the VE/VCO2 slope; Test type: Superiority or Other; p = 0.034, t-test, 1 sided; Compare between metformin and placebo arm; Mean Difference (Net) = -4.45, Standard Deviation 10.72

ADVERSE EVENTS:
Arm/Group | Metformin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/39 | 1/23
Other Adverse Events (participants affected / at risk) | 18/39 | 3/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=39) | Placebo (N=23)
Acute Coronary Syndrome (Cardiac disorders) | 2 (2) | 0 (0) — 2 patients in the metformin arm had acute coronary syndrome prior to starting on metformin. Therefore, reported as serious adverse event. Causality to metformin: Not related.
Prostate Cancer (Renal and urinary disorders) | 0 (0) | 1 (1) — 1 patient in the placebo arm was diagnosed prostate cancer prior to starting on placebo. Therefore reported as serious adverse event. Causality to event: Not related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=39) | Placebo (N=23)
Diarrhoea (Gastrointestinal disorders) | 18 (18) | 3 (3) — Mild to moderate in severity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes